CLINICAL TRIAL: NCT06695182
Title: the Real-world Data of Risk Factor and Its Prognosis in PREmature Coronary ARtery DIseAse Study (PRE-CARDIA)
Brief Title: the Real-world Data of Risk Factor and Its Prognosis in PREmature Coronary ARtery DIseAse Study
Acronym: PRE-CARDIA
Status: Active, not recruiting | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Collaborators: First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Xiao-dong Zhuang, Professor, First Affiliated Hospital, Sun Yat-Sen University
Other Study IDs: PRE-CARDIA study
Record Dates: First submitted 2024-11-05; First posted 2024-11-19 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Premature Coronary Heart Disease
Keywords: Premature coronary heart disease; Risk factor; aging
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- premature coronary artery disease
  Interventions: Behavioral: physical activity

INTERVENTIONS:
Behavioral: physical activity

SUMMARY:
The goal of this observational study is to explore the relationship between biological aging and long-term prognosis of patients with metabolic cardiovascular disease in premature coronary artery disease. The main question[s] it aims to answer [is/are]:

1. Do patients with premature coronary heart disease have accelerated biological aging?
2. What is the prognosis of accelerated biological aging in patients with premature coronary heart disease?

ELIGIBILITY:
Inclusion Criteria:

* Male or female inpatients over 18 years old in the Department of Cardiovascular Medicine;
* Patients with one of the following metabolic cardiovascular diseases [17]: including diabetes, hypertension, coronary heart disease, heart failure, cerebral infarction, dyslipidemia, obesity and hyperuricemia;
* Those who have corresponding inspection data so as to be able to calculate the biological age;
* Obtaining oral informed consent or signing an informed consent form;

Exclusion Criteria:

·NA

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The definition of premature coronary heart disease is that the onset of coronary heart disease in men is ≤55 years old and that in women is ≤65 years old.
Study Population: This study adopts a single-center, one-arm and historical prospective cohort design, and plans to retrospectively collect the data of patients with metabolic cardiovascular diseases hospitalized in the Department of Cardiovascular Medicine of the First Affiliated Hospital of Sun Yat-sen University from January 2013 to now through the electronic medical record system.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
International physical activity questionnaire | Baseline.
  The duration and form of exercise (low, moderate and high intensity) was reported in the form of recall, with higher scores representing more exercise.
Accelerometer | Up to 8 weeks.
  Record participants' daily exercise, more objective than questionnaires.
Cardiopulmonary test | Up to 8 weeks.
  Representation of extreme and sub-extreme motion.
Glucose | Up to 8 weeks.
  Measurement of fasting blood glucose levels to evaluate changes in glucose metabolism and glycemic control. Fasting blood samples are collected in the morning following an 8- to 12-hour fast. Blood glucose concentration is measured in milligrams per deciliter (mg/dL) using a standardized laboratory analyzer to ensure accuracy and consistency.
Hemoglobin A1c (HbA1c) | Up to 8 weeks.
  Measurement of Hemoglobin A1c (HbA1c) levels to evaluate long-term glycemic control over the past 2-3 months. HbA1c is measured as a percentage using a high-performance liquid chromatography (HPLC) method, providing an indication of average blood glucose levels.
Serum creatinine | Up to 8 weeks.
  Measurement of serum creatinine levels to assess renal function and monitor potential changes over time. Serum creatinine is measured in milligrams per deciliter (mg/dL) using an enzymatic assay in a certified laboratory. This measurement serves as a key indicator of kidney function and is used to calculate the estimated glomerular filtration rate (eGFR) as an additional marker of renal health.
Lipid | Up to 8 weeks.
  Measurement of lipid profile, including total cholesterol, low-density lipoprotein cholesterol (LDL-C), high-density lipoprotein cholesterol (HDL-C), and triglycerides, to evaluate cardiovascular risk and lipid metabolism. Fasting blood samples are collected after an 8- to 12-hour fast and analyzed in a certified laboratory using enzymatic colorimetric assays. Results are expressed in milligrams per deciliter (mg/dL).
Serum uric acid | Up to 8 weeks.
  Measurement of serum uric acid levels to assess purine metabolism and monitor for potential hyperuricemia. Serum uric acid is measured in milligrams per deciliter (mg/dL) using an enzymatic colorimetric method in a certified laboratory. This measure provides insight into kidney function and potential risk of gout.
Blood urea nitrogen | Up to 8 weeks.
  Measurement of blood urea nitrogen (BUN) levels to evaluate kidney function and protein metabolism. BUN is measured in milligrams per deciliter (mg/dL) using an enzymatic assay in a certified laboratory, offering an indicator of renal health and nitrogen balance.

SECONDARY OUTCOMES:
Center for Epidemiologic Studies Depression Scale (CES-D) | Up to 8 weeks.
  Assessment of depressive symptoms using the Center for Epidemiologic Studies Depression Scale (CES-D), a validated 20-item self-report questionnaire that measures the frequency of depressive symptoms experienced in the past week. Each item is scored on a 4-point Likert scale, ranging from 0 (rarely or none of the time) to 3 (most or all of the time), with a total score range of 0-60. Higher scores indicate more severe depressive symptoms.
uroQol 5-Dimension 5-Level (EQ-5D-5L) | Up to 8 weeks.
  Assessment of health-related quality of life using the EuroQol 5-Dimension 5-Level (EQ-5D-5L) questionnaire. This tool measures five dimensions of health: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has five response levels, ranging from no problems to extreme problems, resulting in a single health state index score. Additionally, participants provide a self-rated health score on a visual analog scale (VAS) from 0 (worst imaginable health) to 100 (best imaginable health). Higher scores indicate better health-related quality of life.
Multidimensional Sports Self-efficacy Scale (MSES) | Up to 8 weeks.
  Assessment of sports-related self-efficacy using the Multidimensional Sports Self-efficacy Scale (MSES), a validated questionnaire measuring an individual's confidence in performing various aspects of sports performance. The MSES includes subscales for different dimensions, such as physical skill, self-regulation, and coping with pressure. Each item is rated on a Likert scale from 1 (not at all confident) to 7 (extremely confident), with higher scores indicating greater self-efficacy in sports-related skills and resilience.
Chinese self-efficacy for exercise scale (SEE-C) | Up to 8 weeks.
  Assessment of self-efficacy for exercise using the Chinese Self-Efficacy for Exercise Scale (SEE-C), a validated questionnaire designed to measure an individual's confidence in their ability to engage in and sustain exercise. The SEE-C consists of several items that assess self-efficacy across various domains such as initiation, maintenance, and overcoming barriers to exercise. Each item is rated on a Likert scale from 1 (not at all confident) to 5 (extremely confident), with higher scores reflecting greater confidence in one's ability to engage in regular physical activity.